CLINICAL TRIAL: NCT02944344
Title: Four Conversations Randomized Controlled Trial
Brief Title: Four Conversations RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke Cancer Institute (Other); National Comprehensive Cancer Network (Network); Pfizer (Industry); Pillars4Life, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00070790
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage 4; metastatic; hospice; palliative care; end of life; advance directive; oncology; caregiver; provider; coping; support; online
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Death; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Four Conversations Intervention (Experimental): Subjects in this arm will participate in Reimagine's online Four Conversations program during the initial study period of four weeks.
  Interventions: Behavioral: Four Conversations
- Waitlisted Control (Other): Subjects in this arm will continue to receive standard care from their healthcare providers during the initial study period (i.e. no intervention). After four weeks, subjects will then participate in Reimagine's online Four Conversations program.
  Interventions: Behavioral: Four Conversations

INTERVENTIONS:
Behavioral: Four Conversations — The online Four Conversations program consists of tutorial videos, printable documents, and live sessions with a counselor to educate subjects on shared decision making and care planning for those with advanced disease.

SUMMARY:
The purpose of this study is to see whether patients with metastatic breast cancer, their caregivers, and their healthcare providers can improve in shared decision making (SDM) and preparedness around end of life (EOL) planning through participation in Reimagine's online Four Conversations™ program. The goal is to close clinical practice gaps and enhance the quality of care for patients with metastatic breast cancer through increased competence and performance of healthcare providers and healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic breast cancer (MBC), caregiver to patient with MBC who is enrolled in this study, or MBC provider
* Age ≥ 18 years
* Internet access through a computer, laptop, tablet, or other mobile device
* Able/willing to have an online interaction with a Reimagine Pillar Guide
* Providing informed consent
* Able to read/write English

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2018-10-21 (Actual)

PRIMARY OUTCOMES:
Change in patient/caregiver and provider preparedness for decision making as measured by the Preparation for Decision Making Scale | Baseline, Week 4 (waitlisted control only), Post-Intervention (Week 4 or 8)
  The Preparation for Decision Making Scale is a reliable and validated self-reported measure of the patient/caregiver or provider's perception of how useful a decision support intervention is in preparing the respondent to communicate with others making a health decision. Items are summed and scored, then divided by 10; scores can be converted to a 0-100 scale. Higher scores indicate higher perceived level of preparation for decision making.
Change in patient/caregiver decision making self-efficacy as measured by the Decision Self-efficacy Scale | Baseline, Week 4 (waitlisted control only), Post-Intervention (Week 4 or 8)
  The Decision Self-efficacy Scale is a reliable and validated instrument that measures self-confidence or belief in one's abilities in decision making, including shared decision making (SDM). Items are summed, divided by 11, and multiplied by 25. Scores range from 0 to 100 (very confident).
Change in patient self-conflict as measured by the Decisional Conflict Scale | Baseline, Week 4 (waitlisted control only), Post-Intervention (Week 4 or 8)
  The Decisional Conflict scale is a reliable and validated measure of the state of uncertainty about a course of action. Items are summed, divided by 16, and multiplied by 25. Scores range from 0 to 100 (high decisional conflict).

SECONDARY OUTCOMES:
Change in provider end of life (EOL) care knowledge as measured by revised City of Hope EOL Knowledge Assessment | Baseline, Post-Intervention (Week 4)
  The content of the City of Hope End of Life Knowledge Assessment was revised to reflect the program curriculum. Correctly answered questions will be awarded one point, summed, and a total score generated.
Change in patient and caregiver quality of life (QOL) as measured by the PROMIS Global Scale | Baseline, Week 4 (waitlisted control only), Post-Intervention (Week 4 or 8)
  The PROMIS Global Scale is a reliable and validated measure of general perceptions of health. Items are predictive of care utilization and mortality. The scale produces two health scores: physical and mental. Items are summed and converted to t-scores.
Change in patient/caregiver and provider end of life (EOL) conversations as measured by EOL Conversations | Baseline, Week 4 (waitlisted control only), Post-Intervention (Week 4 or 8)
  The EOL Conversations are author-developed questionnaires incorporating items from the Survey on Advanced Care Planning Conversations. Points are totaled and summed.

OTHER OUTCOMES:
Feasibility as measured by completion of advance directive documents | Post-Intervention (Week 4 or 8)
Feasibility as measured by the patient's completion of Reimagine's Worries to Wishes Treatment Plan | Post-Intervention (Week 4 or 8)
Feasibility as measured by Reimagine's Four Conversations program usage, as measured by clickstream data from Reimagine's website and Reimagine staff report | Intervention period (4 weeks)
  Clickstream data associated with viewing videos and other web content (e.g., social community) on the Reimagine website will be collected and analyzed through a web analytics software package. Session attendance will be collected by the Reimagine staff (specially trained counselors called Pillar Guides) and sent to the study team for analysis following each of the online meetings.
Feasibility as measured by satisfaction with Reimagine's Four Conversations program, as measured by the Program Satisfaction & Evaluation questionnaire | Post-Intervention (Week 4 or 8)
  The Program Satisfaction & Evaluation questionnaire was developed by the study team to assess perceived helpfulness of the program in terms of outcomes and patient-provider communication. Points are totaled and summed.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia K Smith, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ryan RE, Connolly M, Bradford NK, Henderson S, Herbert A, Schonfeld L, Young J, Bothroyd JI, Henderson A. Interventions for interpersonal communication about end of life care between health practitioners and affected people. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD013116. doi: 10.1002/14651858.CD013116.pub2. PMID 35802350
- [Derived] Smith SK, Westbrook K, MacDermott K, Amarasekara S, LeBlanc M, Pan W. Four Conversations: A Randomized Controlled Trial of an Online, Personalized Coping and Decision Aid for Metastatic Breast Cancer Patients. J Palliat Med. 2020 Mar;23(3):353-358. doi: 10.1089/jpm.2019.0234. Epub 2019 Oct 22. PMID 31638448